CLINICAL TRIAL: NCT06168526
Title: Acute Effects of Physical Activity on Cognition and Well-being in University Students: ActClass4Brain Project
Brief Title: Acute Effects of Physical Activity on Cognition and Well-being in University Students
Acronym: ActClass4Brain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, Maria Reyes Beltran Valls, Associate Professor, Universitat Jaume I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UJI-B2022-37; CIGE/2021/053 (Other Grant/Funding Number: Generalitat Valenciana)
Record Dates: First submitted 2023-11-22; First posted 2023-12-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Change; Well-Being, Psychological
Keywords: Young adults; Acute physical activity; Attention; Positive affect; Negative affect
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study will be carried out following a crossover design with comparisons between the subjects, in which the cognition and the affective dimensions will be analysed before and after each experimental condition (acute exercise vs. sedentary control).
Masking Description: The assignment to the different conditions will be carried out using a random number generation program stratifying by sex (i.e., the randomizer.org tool).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute physical activity (Experimental): The participants in the experimental activity groups will perform an interval physical activity of different intensity for 16 minutes. The intensity will be controlled during the test by the monitorization of their heart rate using a heart rate monitor. Subsequently, participants will perform an active break in the classroom after finishing one of their usual theory sessions at the intensity of physical activity that proves to have the greatest benefits for cognition and well-being.
  Interventions: Behavioral: Acute physical activity

INTERVENTIONS:
Behavioral: Acute physical activity — Regarding the first aim, participants will go through five different conditions using a within-participants cross-over design in a randomized order: control group (quietly sitting), light intensity (40% VO2max), moderate intensity (63% VO2max), or vigorous intensity (100% VO2max) exercise. All conditions will last 16 minutes and 15 seconds. The exercise conditions will be organized following an interval protocol, which includes 22 bouts of 30 seconds running at the established intensity with 15 seconds of passive rest between bouts. In addition, to achieve the second aim, the active break will be designed taking into account the intensity of physical activity that proves to have the greatest benefits on cognition and well-being.

SUMMARY:
Previous studies in young adults have shown that physical activity can generate positive emotions and improve attention, among other cognitive functions. This highlights the importance of evaluating how physical activity can affect cognition and affective dimensions. However, to date, the dose of physical activity that could be most effective for these variables has not been established. This project aims to study the impact of acute physical activity on brain health in a university setting. Thus, this study will contribute to expand the current scientific literature on the acute effect of physical activity, a topic of great importance both in the educational field and from a public health point of view.

DETAILED DESCRIPTION:
Students in the university stage face many changes in their lives. These changes, partly derived from academic activity, can cause alterations in their lifestyle and brain health (i.e., cognitive, emotional, and behavioural functioning). Due to the negative association of several indicators of brain health with academic performance during the university stage, it is of interest to promote strategies that can favour it. Among them, previous studies in young adults have shown that physical activity can generate positive emotions and improve attention, among other cognitive functions. However, to date, the dose of physical activity (i.e., type, duration, and intensity) that could be most effective for these variables has not been established. Furthermore, previous studies in the matter have been carried out in laboratories and few investigations have analysed outside them the impact of acute physical activity on brain health in university classrooms. Therefore, expanding the current scientific literature on the acute effect of physical activity is of great importance in the educational field, since it would contribute to the design of active proposals aimed at improving brain health with positive implications for students' academic performance and quality of life.

Accordingly, this project aims to carry out an acute physical activity intervention with different intensities and active breaks with students from the Jaume I University (Castellon de la Plana, Spain). More precisely, a total of 210 students between 18 and 24 years old will participate in the intervention.

To achieve it, a randomized crossover study design will be carried out with the groups of participants compensated in terms of number and sex. Attention will be assessed using the d2-R questionnaire and emotional well-being will be assessed using the Positive and Negative Affect Schedule questionnaire. The tests evaluating attention and emotional well-being will be carried out before and after each condition. The experimental conditions will be: control group (quietly sitting), light intensity (40% VO2max), moderate intensity (63% VO2max), or vigorous intensity (100% VO2max) exercise, all lasting 16 minutes. In addition, an active break will be performed at the intensity of physical activity that proves to have the greatest benefits on cognition and well-being.

Taking into account that the lifestyle of students is mainly characterized by the accumulation of prolonged periods of sedentary activity, introducing physical activity in the classroom represents an interesting opportunity for intervention from both an educational and a public health point of view.

ELIGIBILITY:
Inclusion Criteria:

* Not to be diagnosed with psychological and/or cognitive alterations or pathologies that may limit the understanding and following of the instructions provided by another person.
* Not to suffer physical alterations that may limit the practice of physical activity.
* To be between 18 and 24 years old.

Exclusion Criteria:

* To be diagnosed with psychological and/or cognitive alterations or pathologies that may limit the understanding and following of the instructions provided by another person.
* To suffer physical alterations that may limit the practice of physical activity.
* Not to be between 18 and 24 years old.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Attention (cognition) | 10 minutes before and 10 minutes after the intervention protocol
  The participants will take the d2-R test to measure their attention. The test shows different rows of randomly mixed letters from which the target symbol is a "d" with two dashes. The participants must select all the "d" with two dashes while ignoring all the other symbols.
Positive and negative affect (wellbeing) | 10 minutes before and 10 minutes after intervention protocol
  In order to assess the positive and negative affect, the participants will take the Positive and Negative Affect Schedule (PANAS). It is a self-report measure that is made up of two mood scales, one measuring positive affect (the scores ranging from 10 to 50, with higher scores meaning better wellbeing) and the other measuring negative affect (the scores ranging from 10 to 50, with higher scores meaning worse wellbeing).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Reyes Beltran Valls, PhD, Principal Investigator — Universitat Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No
The sharing of the data of the participants in the study with third parties is not foreseen or planned.

REFERENCES:
- [Background] Chan JSY, Liu G, Liang D, Deng K, Wu J, Yan JH. Special Issue - Therapeutic Benefits of Physical Activity for Mood: A Systematic Review on the Effects of Exercise Intensity, Duration, and Modality. J Psychol. 2019;153(1):102-125. doi: 10.1080/00223980.2018.1470487. Epub 2018 Oct 15. PMID 30321106
- [Background] Diener E. Subjective well-being. Psychol Bull. 1984 May;95(3):542-75. No abstract available. PMID 6399758
- [Background] Schmitt A, Upadhyay N, Martin JA, Rojas S, Struder HK, Boecker H. Modulation of Distinct Intrinsic Resting State Brain Networks by Acute Exercise Bouts of Differing Intensity. Brain Plast. 2019 Dec 26;5(1):39-55. doi: 10.3233/BPL-190081. PMID 31970059
- [Background] Leger L, Boucher R. An indirect continuous running multistage field test: the Universite de Montreal track test. Can J Appl Sport Sci. 1980 Jun;5(2):77-84. PMID 7389053
- [Background] Ludyga S, Ishihara T, Kamijo K. The Nervous System as a Pathway for Exercise to Improve Social Cognition. Exerc Sport Sci Rev. 2022 Oct 1;50(4):203-212. doi: 10.1249/JES.0000000000000300. Epub 2022 Jun 24. PMID 35749761
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Erickson KI, Hillman C, Stillman CM, Ballard RM, Bloodgood B, Conroy DE, Macko R, Marquez DX, Petruzzello SJ, Powell KE; FOR 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Physical Activity, Cognition, and Brain Outcomes: A Review of the 2018 Physical Activity Guidelines. Med Sci Sports Exerc. 2019 Jun;51(6):1242-1251. doi: 10.1249/MSS.0000000000001936. PMID 31095081
- [Background] Ludyga S, Gerber M, Brand S, Holsboer-Trachsler E, Puhse U. Acute effects of moderate aerobic exercise on specific aspects of executive function in different age and fitness groups: A meta-analysis. Psychophysiology. 2016 Nov;53(11):1611-1626. doi: 10.1111/psyp.12736. Epub 2016 Aug 24. PMID 27556572
- [Background] Brickenkamp, R., Schmidt-Atzert, L., & Liepmann, D. d2-R. Test de Atención - Revisado. TEA Ediciones. 2022.